CLINICAL TRIAL: NCT00755547
Title: Physical Activity for Overweight Youth at Risk for Type 2 Diabetes Mellitus (POWER) Trial
Brief Title: A Study of the Effects of Exercise Intensity on Insulin Sensitivity in Overweight Youth
Acronym: POWER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Institute of Child Health (Industry)
Responsible Party: Principal Investigator, Jon McGavock, Associate Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SC-5-08-2489-JM; GRT2008-10
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Type 2 Diabetes Mellitus; Adolescent Obesity
Keywords: Childhood; insulin sensitivity; steatosis, spectroscopy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pediatric Obesity; Insulin Resistance; Fatty Liver

ARMS (3):
- High Intensity (Experimental): 70-85% of peak oxygen uptake for 30 min 3-5 days/week.
  Interventions: Other: Aerobic Exercise Training
- Low Intensity (Experimental): 40-55% of peak oxygen uptake for 60 min 3-5 days/week
  Interventions: Other: Aerobic Exercise Training
- Sedentary Control (No Intervention): Regular activities of daily living for 6 months

INTERVENTIONS:
Other: Aerobic Exercise Training — All sessions will be designed to elicit a certain degree of energy expenditure that will progressively increase throughout the trial. Adolescents randomized to the vigorous activity group will perform interval sessions that ensure an average heart rate between 70 and 85% of maximal heart rate reserve while those randomized will perform aerobic activity between 40 and 50% of heart rate reserve. The goal for the trial will be to expend a minimum of 350 kcal. The type of exercise will depend on the preference of each participant however, during the supervised sessions walking/jogging on a treadmill or outdoors will be used to elicit exercise intensities. The three activity sessions held at the YMCA-YWCA facilities in Winnipeg and be supervised by a trained kinesiologist who will record heart rate and perceived exertion for each session.
  Arms: High Intensity; Low Intensity

SUMMARY:
Background:

The investigators know that exercise helps children develop strong bones and muscles and generally stay healthy. What is unclear however, is how much exercise a child needs to lower their risk of developing type 2 diabetes.

Objective:

The investigators will try to find out whether high-intensity exercise for a short-period of time is better than moderately intense exercise for improving the diabetes risk profile in teens who are at risk for type 2 diabetes.

The working hypothesis is that exercise-mediated improvements in insulin sensitivity (a risk factor for diabetes) will be greater following vigorous intermittent physical activity than following low intensity physical activity in overweight adolescents 13-18 yrs at risk for T2DM.

Brief Description of Research Project: Teenagers between the ages of 13 and 18 yrs, who are at risk for type 2 diabetes (either by their family history or an abnormal response to sugar) will be randomly assigned to one of two activity groups or a control group. The activity groups will have supervised exercise sessions 3 to 5 days per week for 6 months. One group will do high-intensity exercise, and the other will do lower-intensity exercise. We will measure how sensitive their body is to insulin and the amount of fat in their muscle and liver tissue at the beginning and end of the exercise intervention.

DETAILED DESCRIPTION:
The Physical activity for OverWEight youth at Risk for type 2 diabetes (POWER) Trial is a randomized controlled clinical trial designed to study the effects of aerobic exercise training regimens differing in intensity (relative to peak fitness) on insulin sensitivity in overweight youth. Additionally, this trial will explore the biologic mechanisms through which chronic physical activity alters lipid metabolism to result in improvements in insulin sensitivity.

We will recruit 90 eligible adolescents and randomly assign them to one of two six-month intervention arms that differ by intensity but elicit similar amounts of energy expenditure: (1) a low intensity continuous activity arm (40-55% of peak oxygen uptake for 60 min); (2) vigorous intensity intermittent activity arm (70-85% of peak oxygen uptake for 30 min) or a sedentary control group. The primary outcome measure of this trial will be insulin sensitivity, measured directly from Bergman's frequently sampled intravenous glucose tolerance test.

ELIGIBILITY:
Inclusion criteria:

* Ethnic minority considered at risk for T2DM
* In utero exposure to hyperglycemia (i.e. mother with gestational or frank diabetes during pregnancy) and/or evidence of hepatic steatosis (serum ALT > 60U/L, ultrasound or MRI-based evidence of steatosis).

Exclusion criteria:

* The investigators will exclude any patients that may have altered insulin sensitivity or tissue lipid content that would confound (mask) the effects of the intervention.
* These include overweight adolescents who:

  * are diagnosed with impaired glucose tolerance or type 2 diabetes
  * are currently being treated with corticosteroids or atypical antipsychotics, as these agents significantly influence carbohydrate metabolism
  * are undergoing puberty (Tanner Stage 2-4) at the time of the investigation, as it is associated with transient changes in insulin sensitivity
  * have an orthopaedic injury that would prevent them from performing the intervention
  * have experienced weight loss or enrolled in weight loss program in the six months prior to the study
  * have a history of alcoholism or drug abuse.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2008-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity measured from Bergman's frequently sampled intravenous glucose tolerance test | 6 months

SECONDARY OUTCOMES:
1H-Magnetic resonance spectroscopy-derived measure of lipid content in liver and muscle tissue | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M McGavock, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Manitoba Institute of Child Health, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Hrubeniuk TJ, Hay JL, MacIntosh AC, Wicklow B, Wittmeier K, McGavock JM, Senechal M. Interindividual variation in cardiometabolic health outcomes following 6 months of endurance training in youth at risk of type 2 diabetes mellitus. Appl Physiol Nutr Metab. 2021 Jul;46(7):727-734. doi: 10.1139/apnm-2020-0707. Epub 2021 Feb 5. PMID 33544653
- [Derived] Mollard RC, Senechal M, MacIntosh AC, Hay J, Wicklow BA, Wittmeier KD, Sellers EA, Dean HJ, Ryner L, Berard L, McGavock JM. Dietary determinants of hepatic steatosis and visceral adiposity in overweight and obese youth at risk of type 2 diabetes. Am J Clin Nutr. 2014 Apr;99(4):804-12. doi: 10.3945/ajcn.113.079277. Epub 2014 Feb 12. PMID 24522441